CLINICAL TRIAL: NCT06923215
Title: The Role of Estimated Glucose Disposal Rate as a Metric for Detection of Metabolic Associated Fatty Liver Disease and Its Severity in Patients With Metabolic Syndrome.
Brief Title: Glucose Disposal Rate as a Metric for Detection of Metabolic Associated Fatty Liver
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira William Ayad Makar, resident at the tropical medicine and gastroenterology in Assuit university., Assiut University
Other Study IDs: Glucose Disposal Rate in MAFLD
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: MAFLD
Keywords: MAFLD; eGDR; Fibroscan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults with suspected/confirmed metabolic syndrome: Adults (18-65 years) with suspected/confirmed metabolic syndrome (IDF criteria) attending a metabolic clinic in Egypt over 12 months. Exclusions include other liver diseases, high alcohol intake, pregnancy, or advanced cirrhosis.

SUMMARY:
A 12-month prospective observational cohort study assessing eGDR's utility in diagnosing MAFLD (via FibroScan® CAP ≥248 dB/m) and correlating it with steatosis/fibrosis severity. Secondary aims compare eGDR to FLI/FIB-4 scores and identify optimal diagnostic cut-offs

DETAILED DESCRIPTION:
Primary Aim

Determine eGDR's diagnostic accuracy for MAFLD using FibroScan® (CAP ≥248 dB/m) as the gold standard.

Secondary Aims

Correlate eGDR with MAFLD severity (steatosis via CAP, fibrosis via liver stiffness measurement [LSM]).

Compare eGDR's performance to Fatty Liver Index (FLI) and FIB-4 in detecting MAFLD and predicting fibrosis.

Identify optimal eGDR cut-offs for MAFLD detection (<6 mg/kg/min) and advanced fibrosis staging (<4 mg/kg/min).

Evaluate eGDR's reclassification improvement (net reclassification index >10%) over existing scores.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* Suspected/confirmed MS per IDF criteria:
* Central obesity (waist circumference ≥94 cm [men]/≥80 cm [women]) plus ≥2 of: Triglycerides ≥150 mg/dL.

HDL <40 mg/dL (men)/<50 mg/dL (women). Blood pressure ≥130/85 mmHg or antihypertensive treatment. Fasting glucose ≥100 mg/dL or diabetes diagnosis.

Exclusion Criteria:

* Other liver diseases (viral/autoimmune hepatitis).

Alcohol intake >20 g/day (men) or >10 g/day (women).

Pregnancy, malignancy, advanced cirrhosis.

Medications affecting metabolism (e.g., steroids)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (18-65 years) with suspected/confirmed metabolic syndrome (IDF criteria) attending a metabolic clinic in Egypt over 12 months. Exclusions include other liver diseases, high alcohol intake, pregnancy, or advanced cirrhosis. All participants undergo:
  Clinical/laboratory assessment: Anthropometrics, blood pressure, fasting glucose, HbA1c, lipid profile, liver enzymes, platelet count.
  eGDR calculation: Formula incorporating waist circumference, hypertension status, and HbA1c.
  FibroScan® evaluation: CAP for steatosis grading (S0-S3) and LSM for fibrosis staging (F0-F4).
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
eGDR will demonstrate high accuracy for MAFLD detection | 3 months
  eGDR will demonstrate ≥0.75 AUC for MAFLD detection and eGDR will show superior specificity compared to FLI/FIB-4.

IPD SHARING:
Plan to Share IPD: No